CLINICAL TRIAL: NCT03215667
Title: Ridge Preservation With Hardening Calcium Phosphate Bone Substitutes and Resorbable Membrane for Implant Site Development on Non-containable Extraction Sites: A Clinical and Histological Prospective Case Series in Humans
Brief Title: Ridge Preservation With Moldable Beta-tricalcium Phosphate Bone Substitute on Non-containable Non-Molar Extraction Sites
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Sunstar Americas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-2016-11-07-1
Record Dates: First submitted 2017-07-10; First posted 2017-07-12 (Actual); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Alveolar Ridge Preservation; Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Device treatment (Experimental): easy-graft CLASSIC (beta-Tricalcium Phosphate) grafting covered with polylactide membrane
  Interventions: Device: easy-graft CLASSIC (beta-Tricalcium Phosphate)

INTERVENTIONS:
Device: easy-graft CLASSIC (beta-Tricalcium Phosphate) — easy-graft will be grafted to a single extraction socket and covered by polylactide membrane to facilitate regeneration of new bone in order to preserve alveolar ridge dimensions.
  Other Names: GUIDOR Bioresorbable Matrix Barrier

SUMMARY:
Purpose of the single arm study is to clinically and histologically evaluate alloplastic in-situ hardening, moldable beta-tricalcium phosphate(TCP) bone graft material and polylactide membrane in alveolar ridge preservation following extraction of non-molar teeth with non-containable extraction sockets.

ELIGIBILITY:
Inclusion Criteria:

* adequate restorative space for a dental implant restoration, if the subject decides previous to study participation that they would like an implant. Note, agreement to implant placement is not a requirement of the study
* minimum of 10-mm vertical bone without impinging on adjacent vital structures (Maxillary sinus, neurovascular bundles)
* single-rooted tooth to be extracted
* American Society of Anesthesiologists (ASA) Physical Status Classification I or II
* age >18 years old
* subjects who had >50% of height on any portion on the buccal wall of dehiscence and/or fenestration of the extraction socket following extraction will be included from this study
* adjacent teeth to extraction site will be present during healing period
* willingly sign informed consent and authorization.

Exclusion Criteria:

* do not meet any inclusion criteria
* pregnancy or nursing woman
* subjects with active systemic or localized infection (exclude chronic periodontitis)
* subjects with a history of any medical conditions that contraindicated or weighed against dental implant placement such as history of bisphosphonate drug use, chemotherapeutic or immunosuppressive agents, autoimmune disease, or poorly controlled diabetes (HBA1c>7%)
* subjects with smoking habit (more than 10 cigarettes per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-11-03 (Actual); Study Completion 2019-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Dentistry, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device Treatment
Started | 9
Completed | 5
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Device Treatment
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Radiographic Measurements of Bone Ridge Dimensions
Description: Cone-beam computed tomography (CBCT) was taken at the ridge preservation procedure (baseline) and 3 months after the procedure. The horizontal ridge width was measured at 1, 3, 5 and 7 mm below the alveolar bone crest. Overall change is the average of all measurements.
Time Frame: Change from Baseline at 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Device Treatment
Number analyzed (Participants) | 5
mm
  Overall | 1.59 (1.05)
  1 mm below the alveolar bone crest | 1.89 (1.03)

2. Secondary Outcome: Change in Digital Measurements of Soft Tissue Dimensions
Description: Pre- and post-surgery casts were made from impressions and scanned with a digital scanner. The soft tissue width was measured at 1, 3 and 5 mm below the ridge crest. Overall change is the average of all measurements.
Time Frame: Change from baseline at 5 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Device Treatment
Number analyzed (Participants) | 5
mm
  Overall | 0.99 (2.18)
  1mm below the ridge crest | 2.57 (1.35)

ADVERSE EVENTS:
Time Frame: 5 months after ridge preservation surgery
Arm/Group | Device Treatment
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT03215667/Prot_SAP_001.pdf